



### Participant Information Sheet

## Pilot study title: Validation and implementation of a Digital Assessment Routing Tool (DART) as an alternative to physiotherapy-led remote triage

# Running title Does an online digital assessment tool called DART work as well as a remote consultation with a physiotherapist for musculoskeletal problems?

#### Researcher's name

Mr. Harry Hanuman Sing Research Assistant Centre for Sport and Exercise Medicine Mile End Hospital, London E1 4DG h.h.sing@qmul.ac.uk Ms. Cabella Lowe PhD student Centre for Sport and Exercise Medicine Mile End Hospital, London E1 4DG c.lowe@qmul.ac.uk

#### **Queen Mary Ethics of Research Committee reference number:**

#### Invitation

We would like to invite you to be part of this research project. You should only agree to take part if you wish to do so; it is entirely up to you. If you choose to not take part, there won't be any disadvantages for you, and you will hear no more about it.

Please take time to read the following information carefully before you decide whether or not to take part. This will tell you why the research is being done and what you will be asked to do should you agree to take part. Please ask if there is anything that is not clear or if you would like more information.

#### What is the purpose of the study and what would taking part involve?

One in five people in the United Kingdom suffers from a problem with their joints, muscles or other soft tissues. For these people, getting help quickly means getting better faster. Some treatments like physiotherapy or a self-help programme can help, but it can take a while to get to the right person who can help you. Some people need to see their GP first or may be asked to speak to a physiotherapist on the phone before they can get the right help.



Our study will explore a new way for people to quickly get the care they need using a system called DART (Digital Assessment Routing Tool). DART is an on-line system you can use on a mobile device or home computer. DART asks a series of questions and will be able to sign-post you to the right type of help for your problem.

If you wish to participate in the study, we will ask you to complete an online assessment of your problem on your mobile phone, tablet, laptop or computer and to complete two short online questionnaires. You will still get an appointment to speak to a physiotherapist and have any treatment you need, regardless of whether you take part in the study or not.

This is the process if you take part:



Your physio telephone or video consultation will be recorded for study-related purposes and may be reviewed by an expert panel. The recording will be kept confidential and only accessible by the research team. It will be deleted at the end of the study. The information about your musculoskeletal problem and other non-identifiable participant information, such



as your age and gender, will be collected and retrieved from DART or Optima Health's electronic patient records. Please note, any of your records, information or data from the NHS will not be accessed or requested in any way. Your information will not be cross-checked with any other source of information.

#### Why am I being invited?

You are being invited to participate in our research study because you are an adult aged 18 years or above who shows signs of a musculoskeletal problem (a problem with the joint, muscle or soft tissue).

#### Do I have to take part?

No, it is up to you to decide whether to take part. If you do decide to take part, you will be given this information sheet to keep and be asked to electronically sign an online written consent form. You can withdraw from the study at any time without needing to provide a reason, and with no disadvantages to your usual care.

#### What are the possible benefits of taking part?

There is no guarantee that this study will benefit you. However, the information we gather from the trial will help us to test and improve DART, which we hope will allow people to access the right treatment quicker. There will be no changes to your treatment by taking part in this study.

#### What are the possible disadvantages and risks of taking part?

We do not anticipate any disadvantages or risks to you from taking part in this research study. The referral process will take slightly longer than usual due to the extra DART assessment. We have carefully planned the study to minimise the extra time required. You will still receive your treatment on the same day as you would do normally.

#### **Expenses and payments**

We do not offer any payment or cover expenses for your participation in this study.

#### What information about me will you be collecting?

We will be collecting the responses you have given to the questions in DART and the on-line questionnaires. The physiotherapist's clinical notes will be stored as usual in Optima Health's electronic patient record, which will only be accessed by a member of the research team. Information important for the study, such as your age and gender, will also be taken from the clinical record. All the study information will be assigned to your study reference number to keep your responses and information confidential.

#### How will my data be stored and who will have access to it?

All electronic information (signed consent form, responses to questionnaires, DART assessment and information from the physiotherapy assessment), will be stored on the central servers of Optima Health and of Queen Mary, University of London.



Your data will be stored in a non-identifiable format. Your name and other identifiable information will be replaced by a unique code. To reduce the risk of disclosure, any personal identifiable data will be stored separately from the research data on the central servers of Optima Health and will only be accessible by the research team.

#### When and how will my data be destroyed?

The retention period of your data will be five years after the study has ended. This is in line with Queen Mary retention schedule and information policy. The data will then be destroyed or archived, but you may always request to have your identifiable data destroyed before this date.

#### How will my data be used and shared?

Your data will be stored in an anonymised format. It will be analysed, and we hope to publish the findings in a peer-reviewed medical or scientific journal.

This study is part of a larger doctoral research project developing DART and you are welcome to ask the study team for the results of the study if you wish.

#### **Queen Mary's privacy notice for research participants**

Please read <u>Queen Mary's privacy notice for research participants</u> containing important information about your personal data and your rights in this respect. If you have any questions relating to data protection, please contact Queen Mary's Data Protection Officer, Queens' Building, Mile End Road, London, E1 4NS or data-protection@gmul.ac.uk or 020 7882 7596.

#### What will happen if I want to withdraw from this study?

You have the right to withdraw at any time during the study without providing a reason for it. This will not have any disadvantages for you in any way. If you do withdraw, identifiable data will be destroyed securely in accordance with the UK Policy Framework for Health and Social Care research; however, data that is already anonymised or coded for analysis will not be changed.

#### What should I do if I have any questions or concerns about this study?

If you have any questions or concerns about the manner in which the study was conducted please, in the first instance, contact the researcher(s) responsible for the study. If you have a complaint which you feel you cannot discuss with the researchers then you should contact the Research Ethics Facilitators at <a href="mailto:research-ethics@qmul.ac.uk">research-ethics@qmul.ac.uk</a> or Queen Mary Ethics of Research Committee, Room W104, Queens' Building, Mile End Campus, Mile End Road, London, E1 4N or Queen Mary Ethics of Research Committee, Joint Research Management Office (JRMO) Empire House, 65 - 75 New Road, Whitechapel, London, E1 1HH. When contacting the Research Ethics Facilitators, please provide details of the name or description the study or QMERC reference number, the researcher(s) involved, and details of the complaint you wish to make.

#### Contact details



Researchers: Harry Hanuman Sing

Research Assistant h.h.sing@qmul.ac.uk

Centre for Sport and Exercise Medicine Mile End Hospital, London E1 4DG (Optima Health – phone number pending)

Ms. Cabella Lowe PhD student

Centre for Sport and Exercise Medicine Mile End Hospital, London E1 4DG

c.lowe@qmul.ac.uk

(Optima Health – phone number pending)

Supervisor: Professor Dylan Morrissey

Professor of Sport and Musculoskeletal Physiotherapy

Centre for Sport and Exercise Medicine Mile End Hospital, London E1 4DG

d.morrissey@qmul.ac.uk

02082238839